CLINICAL TRIAL: NCT01239108
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study of SGI-1776, a PIM Kinase Inhibitor, in Subjects With Relapsed/Refractory Leukemias
Brief Title: Study of SGI-1776, a PIM Kinase Inhibitor, in Subjects With Relapsed/Refractory Leukemias
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The dose limiting toxicity of cardiac QTc prolongation was identified and demonstrated unsafe to continue clinical development of this molecule.
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-1776-02
Record Dates: First submitted 2010-11-05; First posted 2010-11-11 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Relapsed/Refractory Leukemias
MeSH Terms: conditions — Leukemia | interventions — SGI 1776

INTERVENTIONS:
Drug: SGI-1776 — SGI-1776 will be administered orally at escalating dose levels ranging from 350 to 1600 mg/day based on the dose escalation levels of the ongoing, first-in-human study.

SUMMARY:
Dose escalation study for subjects with Leukemia that has returned or has not responded to standard treatment.

DETAILED DESCRIPTION:
A Phase 1, Multicenter, Open-label, Dose-escalation Study of SGI-1776, a PIM Kinase Inhibitor, in Subjects with Relapsed/Refractory Leukemias

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with a confirmed diagnosis of leukemia unresponsive to curative therapy
2. Eastern Cooperative Oncology Group performance status of 0 to 2
3. Total bilirubin ≤ 1.5 X upper limit of normal (ULN); aspartate transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT) ≤ 3 X ULN; serum creatinine ≤ 2 X ULN
4. Normal cardiac function with left ventricular ejection fraction ≥ 50% at screening
5. No clinically significant abnormalities on screening electrocardiogram (ie, QTc interval must be < 470 msec for women and < 450 msec for men and no history of torsades de pointes)
6. No reproductive potential or willing to use 2 methods of contraception during the study and for 30 days after the last dose
7. Able to understand the purpose and risks of the study and provide informed consent and authorization to use protected health information

Exclusion Criteria:

1. A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of oral SGI-1776, or put the study outcomes at undue risk
2. Significant cardiovascular disease
3. Malabsorption syndrome
4. Symptomatic central nervous system metastases or lesions for which treatment is required
5. Received prior radiation therapy within 4 weeks of first dose
6. Grade ≥ 2 toxicity (other than alopecia) continuing from prior anticancer therapy including radiation
7. Treatment with any investigational drug within 3 weeks of the first dose
8. Use of systemic corticosteroids (other than for premedications or intermittent doses such as those used for allergic reactions and control of asthma) or myelosuppressive chemotherapy within 2 weeks of the first dose treatment with nitrosoureas or mitomycin C within 3 weeks of the first dose of SGI 1776
9. Uncontrolled active systemic infections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The MTD as determined by the incidence of DLTs in the first 4 weeks of each dosing cohort | July 2011

SECONDARY OUTCOMES:
• Frequency, severity, and relationship of adverse events (AEs) and serious adverse events (SAEs) • | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States